CLINICAL TRIAL: NCT03709043
Title: A-HACK Project: Addressing Heavy Alcohol Use Consumption With Kudzu
Brief Title: Addressing Heavy Alcohol Use Consumption With Kudzu
Acronym: A-HACK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenn-Milo Santos (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Glenn-Milo Santos, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-25073; R01AA025930-01A1 (NIH)
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder; Sexually Transmitted Diseases
MeSH Terms: conditions — Alcoholism; Sexually Transmitted Diseases | interventions — Counseling; Ethanol; Urinalysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kudzu (Experimental): Standardized kudzu
  Interventions: Drug: Standardized kudzu; Diagnostic Test: Sexually transmitted infection testing:; Behavioral: Medical Management (MM) counseling for alcohol use:; Diagnostic Test: Urinalysis for novel alcohol biochemical markers for recent alcohol use:; Diagnostic Test: Dried Blood Spot (DBS) Testing for PEth:; Behavioral: Behavioral survey measurements:; Behavioral: Ecological Momentary Assessment procedure:
- Control (Placebo Comparator): Placebo
  Interventions: Other: Placebo; Diagnostic Test: Sexually transmitted infection testing:; Behavioral: Medical Management (MM) counseling for alcohol use:; Diagnostic Test: Urinalysis for novel alcohol biochemical markers for recent alcohol use:; Diagnostic Test: Dried Blood Spot (DBS) Testing for PEth:; Behavioral: Behavioral survey measurements:; Behavioral: Ecological Momentary Assessment procedure:

INTERVENTIONS:
Drug: Standardized kudzu — Standardized kudzu
  Arms: Kudzu
Other: Placebo — Placebo
  Arms: Control
Diagnostic Test: Sexually transmitted infection testing: — At baseline and month 3 visits, all participants will be tested for syphilis (serum RPR), Neisseria gonorrhea and Chlamydia trachomatis (urine, pharyngeal swab, and rectal swab nucleic acid amplification [NAAT]) through an established protocol that has been validated by our Public Health Laboratory (PHL) and others.
Behavioral: Medical Management (MM) counseling for alcohol use: — MM has been used in a targeted pharmacotherapy trial and our team has successfully used MM in AUD trials. MM is a low-intensity supportive program designed to increase problem recognition and enhance motivation to change maladaptive alcohol use patterns. Participants will receive individual 20 minute MM sessions weekly from trained staff supervised by a clinical psychologist.
Diagnostic Test: Urinalysis for novel alcohol biochemical markers for recent alcohol use: — Urine samples will be collected at Enrollment, Month 1, Month 2 and Month 3 visits and tested for ethyl glucuronide (EtG) to determine recent alcohol consumption in the past three days. EtG is a relatively novel, highly sensitive indicator for recent alcohol consumption; this alcohol biomarker is detectable in urine for approximately 72 hours.
Diagnostic Test: Dried Blood Spot (DBS) Testing for PEth: — DBS samples will be collected at enrollment, weeks 12, and post-treatment visits at month 3. Samples will be dried overnight using standardized methods. PEth testing of DBS samples will be conducted at the United States Drug Testing Laboratories in Des Plaines, IL using liquid chromatography-tandem mass spectrometry system following extraction into methanol.
Behavioral: Behavioral survey measurements: — Standardized and validated behavioral measures will be assessed using audio computer administered surveys (ACASI) to minimize underreporting of risk activities and standardize data collection.To minimize potential social desirability bias, staff will not have access to data during the trial.
Behavioral: Ecological Momentary Assessment procedure: — Participants will receive daily SMS texts to collect data on alcohol consumption, number of drinks on drinking days, targeted medication administration prior to anticipated drinking sessions, and sexual risk behaviors

SUMMARY:
Drinking multiple alcoholic drinks on a single occasion (binge drinking), has many negative health risks but interventions to address this behavior remain limited. This double-blind, placebo-controlled randomized clinical trial will test whether kudzu, an herbal supplement, can reduce heavy alcohol use and alcohol-associated sexual behaviors among sexually-active, binge-drinking individuals at high risk for HIV infection.

DETAILED DESCRIPTION:
This study, entitled "The Harness Study" is a double-blind, placebo-controlled, two-arm trial in which 120 binge drinkers with AUD will be randomly assigned to receive 12 weeks of kudzu or placebo, to be taken on an as-needed basis with 1- and 3-month post-treatment follow-up visits. This efficacy study will enroll sexually active, binge drinkers with AUD because they are the most likely population to benefit from this intervention by limiting harms associated with heavy alcohol use and decreasing alcohol-related sexual risk behaviors. A study clinician will perform the Structured Clinical Interview for the DSM-V (SCID) to screen for AUD and determine eligibility. Upon enrollment, 120 participants will be randomized 1:1 to kudzu extract (2 grams) or placebo for targeted administration. Participants will be seen weekly for behavioral surveys, urinalyses, study drug dispensing, and alcohol use counseling. Safety laboratory assessment, vital signs, and the audio computer assisted survey instrument (ACASI) will be completed monthly. Efficacy, tolerability, and acceptability (Specific Aims 1-4) will be assessed upon trial completion as measured by number of binge drinking occasions and numbers of drinks on drinking days via timeline follow-back at weekly visits; number of EtG-positive urine samples; sexual risk behavior data through monthly surveys via ACASI; frequency of adverse events; and cumulative medication adherence data at week 12. Durability of intervention effects will be evaluated at 1- and 3-month post-treatment visits.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported anal or vaginal sex in the prior three months while under the influence of alcohol, or reported missing ART or PrEP due to alcohol use in the prior 3 months;
2. at least one binge-drinking (five or more drinks on a single occasion for men; four or more drinks for women) session per week in the prior three months;
3. having an AUD by DSM-5 SCID criteria (includes hazardous and harmful use);
4. interested in reducing binge alcohol consumption;
5. HIV negative by rapid antibody test and HIV pooled RNA test; or HIV positive with a medical record documentation of HIV infection.* For HIV-positive individuals, having a CD4 cell count >100 cells/mm3 and having suppressed HIV viral load with < 50 copies/mm3; *
6. no current acute illnesses requiring prolonged medical care;
7. no chronic illnesses that are likely to progress clinically during trial participation;
8. able and willing to provide informed consent and adhere to visit schedule;
9. age 18-70 years;
10. baseline CBC, total protein, albumin, glucose, alkaline phosphatase, creatinine, BUN, and electrolytes without clinically significant abnormalities as determined by study clinician in conjunction with symptoms, physical exam, and medical history;

(*Note: Participants newly diagnosed with HIV at screening are eligible for the study but we will postpone their enrollment until they are virally suppressed with HIV viral load < 50 copies/mm .)

Exclusion Criteria:

1. Any psychiatric (e.g., depression with suicidal ideation) or medical condition that would preclude safe participation in the study;
2. known allergy/previous adverse reaction to kudzu;
3. moderate/severe liver disease (AST, ALT > 5 times upper limit of normal);
4. impaired renal function (creatinine clearance < 50 ml/min);
5. currently participating in another intervention research study with potential overlap;
6. current severe substance-use disorder (exclusive of nicotine, cannabis or alcohol) as determined by DSM-V SCID criteria;
7. pregnant women;
8. HIV positive individuals who are not virally suppressed;
9. any condition that, in the principal investigator and/or study clinician's judgment interferes with safe study participation or adherence to study procedures
10. not willing to learn how to send EMA surveys.

(*Note: Eligible participants who have a partner currently in the study will be enrolled and randomized after their partner has completed their in-treatment follow-up, to reduce the concerns of contamination between treatment conditions. Additionally, we will exclude individuals with impaired renal function as a general precaution. Pharmacokinetic data on kudzu is limited. Puerarin is present in the urine of rats for 4-72 hours after oral administration, thus there is renal elimination of the active compound, as well as it's metabolite, equol. For this reason, we prefer to be cautious by limiting enrollment to those with reasonable renal function. We selected eGFR < 50mL/min as that is the level at which most products with renal clearance begin to demonstrate risks of increased toxicity.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
number of binge drinking days | 7 days
  Binge-drinking (five or more drinks on a single occasion for men; four or more drinks for women)

SECONDARY OUTCOMES:
proportion of ethyl glucuronide (EtG) positive urines | 7 days
  Urine samples will be collected weekly and tested for ethyl glucuronide (EtG) to determine recent alcohol consumption in the past three days.

OTHER OUTCOMES:
number of sexual intercourse partners | 30 days
  Self-reported sexual intercourse partners
number of condomless sexual intercourse events | 30 days
  Self-reported of condomless sexual intercourse events
proportion of participants testing positive of sexually transmitted diseases | 30 days
  all participants will be tested for syphilis (serum RPR), Neisseria gonorrhea and Chlamydia trachomatis (urine, pharyngeal swab, and rectal swab nucleic acid amplification at baseline and Month 3 visits

CONTACTS AND LOCATIONS:
Overall Officials: Glenn-Milo Santos, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03709043/Prot_SAP_000.pdf